CLINICAL TRIAL: NCT01100450
Title: Pilot Study to Determine Feasibility, Acceptance, and Efficacy of a 12-week Progressive Resistance Training Exercise Protocol in Patients With Class III Obesity Preparing for Bariatric Surgery.
Brief Title: Progressive Resistance Training in Patients With Class III Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Miguel Alonso-Alonso, MD, Assistant Professor of Surgery, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009P000083
Record Dates: First submitted 2009-10-16; First posted 2010-04-09 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: bariatric surgery; class III obesity; resistance training; strength; fitness
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistance Training (Experimental)
  Interventions: Behavioral: Progressive Resistance Training

INTERVENTIONS:
Behavioral: Progressive Resistance Training — 12-week progressive resistance training (PRT) exercise program

SUMMARY:
To test the strength and physical performance outcomes of a 12-week progressive resistance training (PRT) exercise program in a small cohort of patients with Class III obesity who are preparing for bariatric weight loss surgery at Beth Israel Deaconess. The study will also test patient compliance to the 12 week PRT program. Whereas PRT exercise is currently recommended as a part of preoperative clinical care for bariatric surgery patients, little research has been done to measure the acceptance and effectiveness of a standardized PRT exercise protocol for improving health and perioperative care. Preliminary data from this study could be used to justify larger studies and further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years old
* A BMI of ≥40 kg/m2
* Considering Weight Loss Surgery at BIDMC
* Participating in multidisciplinary preoperative program:

  * been determined by a mental health professional (i.e., psychologist or social worker) to be well-informed, motivated, and not symptomatic for psychopathology that would put the person at risk for injury or failure with WLS
  * expressed strong desire for significant weight loss
  * experienced documented failure of long-term weight loss using nonsurgical methods
  * been informed of and accepts risks of surgery
* Cleared by their primary care physician to be in stable health and capable of moderate level exercise
* Willing to comply with expected attendance and participation at all intervention sessions and testing appointments
* Has reliable transportation to the intervention location

Exclusion Criteria:

* Orthopedic limitations that would preclude exercise testing and training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test | Before training - Week 1
  Subjects are instructed to walk from one end to the other of a 30- meter hallway at their own pace, while attempting to cover as much ground as possible in the allotted 6 minutes. Subjects are allowed to stop and rest during the test, but were instructed to resume walking as soon as they felt able to do so. Total distance walked was recorded at the end of the test.
6-Minute Walk Test | After training - Week 12
  Subjects are instructed to walk from one end to the other of a 30- meter hallway at their own pace, while attempting to cover as much ground as possible in the allotted 6 minutes. Subjects are allowed to stop and rest during the test, but were instructed to resume walking as soon as they felt able to do so. Total distance walked was recorded at the end of the test.

SECONDARY OUTCOMES:
Muscle Fatigability Test | Before training-Week 1
  After appropriate warm-up, subjects performed as many repetitions as possible against a resistance set to 80% or 70% (leg and chest respectively) of their pre-intervention 1-repetition maximum resistance. Fatigability tests measures the ability to sustain a static muscle contraction or make repetitive submaximal dynamic contractions. The test was administered using the leg press and chest press machines (Nautilus Nitro).
1-repetition maximum muscle strength test | Before training-Week 1
  The subject performs repeated single repetitions of leg press and chest press, separated by 60-second rest periods. Resistance is increased systematically at each repetition until the person's maximum voluntary muscle force cannot move the resistance through the full range of motion. The greatest resistance (measured in lbs.) a person can move through a full range of motion is recorded as the "one-repetition maximum." Tests were performed on leg and chest press machines (Nautilus Nitro).
Muscle Fatigability Test | After training-Week 12
  After appropriate warm-up, subjects performed as many repetitions as possible against a resistance set to 80% or 70% (leg and chest respectively) of their pre-intervention 1-repetition maximum resistance. Fatigability tests measures the ability to sustain a static muscle contraction or make repetitive submaximal dynamic contractions. The test was administered using the leg press and chest press machines (Nautilus Nitro).
1-repetition maximum muscle strength test | After training - Week 12
  The subject performs repeated single repetitions of leg press and chest press, separated by 60-second rest periods. Resistance is increased systematically at each repetition until the person's maximum voluntary muscle force cannot move the resistance through the full range of motion. The greatest resistance (measured in lbs.) a person can move through a full range of motion is recorded as the "one-repetition maximum." Tests were performed on leg and chest press machines (Nautilus Nitro).

CONTACTS AND LOCATIONS:
Overall Officials: George L Blackburn, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts